CLINICAL TRIAL: NCT02242604
Title: Phenotypic Characterization of Neuropsychologic and Physical Performance in Geriatric Patients Suffering From Hyponatremia.
Brief Title: Characterization of Neuropsychologic and Physical Performance in Geriatric Patients With Hyponatremia.
Status: Completed | Type: Observational
Sponsor: Volker Burst (Other)
Responsible Party: Sponsor-Investigator, Volker Burst, MD, University of Cologne
Organization: University of Cologne (Other)
Other Study IDs: V1.1; DRKS00005776 (Registry Identifier: DRKS)
Record Dates: First submitted 2014-09-08; First posted 2014-09-17 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Hyponatremia
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Not treatment: Patients with the age of 70 years or above, that have a serum sodium of below 130 mmol/L on admission. All patients will be routinely evaluated at admission with a standardized multidimensional geriatric assessment (MGA) consisting of a battery of validated assays.
  Interventions: Other: Multidimensional Geriatric Assessment (MGA)

INTERVENTIONS:
Other: Multidimensional Geriatric Assessment (MGA) — The MGA contains the following tests:
  1. Barthel Katz Index (activity of daily living, ADL)
  2. Mini Mental State Test (MMST)
  3. DemTec (dementia detection test)
  4. Clock Test
  5. Geriatric Depression Scale (GDS)
  6. Tinetti Test
  7. TUG (timed up-and-go Test)
  8. Esslinger Transfer Scale (ETS)
  9. Handgrip Test
  10. Mini Nutritional Assessment (MNA)

SUMMARY:
Our purpose is to investigate the improvement of the cognitive, neuropsychologic and physical capabilities using a standardized multidimensional geriatric assessment (MGA) consisting of a battery of validated assays after correction of hyponatremia in patients 70 years or older.

DETAILED DESCRIPTION:
With an occurrence of up to 30%, hyponatremia, defined as a serum sodium concentration of less than 135 mmol/L, is the most commonly encountered electrolyte disorder in hospitalized patients today. The highest incidence of hyponatremia is found in the elderly.

Retrospective analyses clearly show an association between hyponatremia and mortality as well as morbidity and this association is not confined only to severely decreased sodium levels. Hyponatremia can be an acute and life-threatening condition, which is usually reflected by severe signs and symptoms, e.g. coma or seizures,but more often it is of chronic nature, and symptoms may be subtle or even apparently absent due to cerebral adaptation processes. Signs and symptoms include, among others, nausea, drowsiness, cognitive impairment, memory deficits, depression, muscle cramps, or gait instability. However, our knowledge of the highly diverse clinical picture of hyponatremia stems from anecdotic reports and experiments that were performed by the investigators on themselves in the 1930ies. Thus, no accurate and thorough description of the symptomatology of hyponatremiain disease has been carried out so far, except maybe for the extreme conditions, i.e. in patients suffering from seizures or coma. This is why especially patients with chronic mild-to-moderate hyponatremia (sometimes defined as a sodium concentration > 125 mmol/L) who may well have subtle or unspecific symptoms are often perceived as being asymptomatic. Recent investigations have demonstrated that such patients have a significantly increased risk for falls and bone fractures and reduced cognitive capacities. Moreover, anecdotic reports have shown that some patients that were believed to suffer from depression or dementia improved markedly after correction of their concomitanthyponatremia. There is also mounting evidence that hyponatremia induces osteoporosis which adds to the risk of bone fractures. Furthermore, in the SALT-trials, the mental component of the SF-12 questionnaire (Short Form-12) improved significantly after hyponatremia had been corrected. Interestingly, the mean sodium concentration prior to treatment was 129 mmol/L indicating mild or moderate hyponatremia. Given the high prevalence of mild-to-moderate hyponatremiain the elderly, unspecific symptoms like mood instability, cognitive deficits or others, thatare often attributed to old age could simply be a consequence of their low sodium level.

To this end, it might well be that by treating hyponatremia the morbidity/mortality in this population could be reduced and quality of life improved. In light of the growing medico-economic challenges we are facing secondary to the steadily increasing life expectancy and the demographic evolution in the western world and the medical problems that come along with this development the influence of successful correction of hyponatremia on mental and physical health should be evaluated. To our knowledge this has not been investigated so far.

The syndrome of inappropriate ADH secretion (SIADH) accounts for more than a third of all cases of hyponatremia and probably is by far the most frequent aetiology of chronic mild to moderate hyponatremia. While newly developed SIADH is often induced by malignancies, pulmonary or cerebral disease in the general population, longstanding chronic hyponatremia in elderly is usually due to idiopathic or drug-associated SIADH. Apart from SIADH, hypovolemia or reduction of the effective arterial blood volume, e.g. in cardiac failure or liver cirrhosis, are common causes of hyponatremia. Although hyponatremia might have an impact on the mental and physical status as well as on the patient's prognosis regardless of the underlying cause, most aetiologies except for SIADH might be confounding factors, since they often induce a "hyponatremia-like" clinical picture by themselves, e.g. hepatic encephalopathy in liver disease etc. Another possible confounder may be hemoglobin. Recent work shows that hyponatremia is associated with anaemia, which is a highly prevalent symptom in elderly patients and an acknowledged risk factor for poor outcome in this population. The underlying pathogenesis of this association is still unknown. Regarding the fact that anaemia and hyponatremia are both risk factors for increased morbidity and mortality in elderly patients that are potentially curable, analysis of influence on the multidimensional geriatric assessment (MGA) before and after correction is challenging. To our knowledge, these possible confounders have not been accounted for in the existing literature. Moreover, no accurate evaluation of the origin of hyponatremia has been reported.

ELIGIBILITY:
Inclusion Criteria:

* age of 70 years or above
* serum sodium of 130 mmol/L and below

Exclusion Criteria:

* patients not capable of giving informed consent
* patients on intensive care unit (ICU)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: A total of 150 patients with the age of 70 years or above, that are admitted to the Department for Geriatric Medicine of the University of Cologne, that have a serum sodium of below 130 mmol/L on admission, and that have complete datasets that allow for unequivocal determination of the etiologic cause of hyponatremia will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of the impact of serum sodium concentration on geriatric assessment scores. | Day of admission - 14 to 21 days
  The impact of serum sodium concentration on geriatric assessment scores will be evaluated individually for each assessment score in a linear model, independent variables being a) increment of serum sodium [mmol/L] from the time of the first MGA at hospital admission to the time of the second MGA prior to discharge, and b) baseline serum sodium [mmol/L] at the time of the first MGA at hospital admission, the dependent variable being change of assessment score. A subgroup analysis will be done for SIADH patients.
  The association between geriatric assessments and serum sodium [mmol/L] will be analysed by correlation analysis at the time of the first and second MGA.

SECONDARY OUTCOMES:
Influence of anaemia as a confounder. | day of admission - 14 to 21 days
  To test for a possible influence of anaemia as a confounder, similar analyses will carried out using haemoglobin [g/dl] as the independent factor and compared to the above mentioned analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, MD, Principal Investigator — Department II of Internal Medicine, Nephrology - University Hospital of Cologne
Locations (1):
- Department for Geriatric Medicine - University of Cologne, Cologne, Germany